CLINICAL TRIAL: NCT01556711
Title: Assessment of Head Injury in the Emergency Department: Clinical Validation of the BrainScope® Ahead™ Technology
Brief Title: Assessment of Head Injury in the Emergency Department Using BrainScope® Ahead® Technology
Acronym: B-AHEAD II
Status: Completed | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: B-AHEAD II Trial
Record Dates: First submitted 2012-03-05; First posted 2012-03-16 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Brain Injuries; Craniocerebral Trauma
Keywords: Head Injury; Head Trauma; TBI (Traumatic Brain Injury); Emergency Department
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Brain Injuries, Traumatic; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Head Injury: Males and females ages 18 to 80 (the entire age range), who are admitted to the ED, who are suspected of a traumatically induced structural brain
- Control: A 'normal' control group will be recruited for comparison and will consist of ED patients ("ED normal control group) who have sustained an injury but do not exhibit any trauma above the clavicle and no history of MVA requiring an ED visit or TBI within the past one (1) year, and no primary complaint of syncope

SUMMARY:
The objectives of the study are to document device performance with respect to the primary and secondary endpoints.

DETAILED DESCRIPTION:
The purpose of the current study is proposed to prospectively validate the BrainScope Ahead® M-100 device design, performance, and labeling with respect to the device's target intended use and indications for use:

* Primary Endpoint:

  * Structural Injury Assessment
  * There are four co-primary endpoints in this study: two sets of sensitivity and specificity to divide the data into three classes.
  * Using a BrainScope classification algorithm, the Ahead® M100 will identify subjects showing sensitivities among 3 classes: Green-normal, nonhead injured controls,Yellow-head injured subjects who do not exhibit brain electrical activity that is consistent with a structural brain injury observable on CT or for whom CT was not deemed necessary,Red-head injured subjects who exhibit brain electrical activity consistent with a structural brain injury observable by CT.
* Secondary Endpoint:

  * Functional Injury Assessment
  * There are two co-secondary endpoints for the secondary objective, the sensitivity and specificity to split Yellow from the primary endpoint into two sub groups depending on degree of brain functional impairment observable by an evaluation of the clinical findings on a clinical charter used as the assessment of truth.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 to 80 (the entire age range), who are admitted to the Emergency Department (ED), who are suspected of a traumatically induced structural brain injury and/or clinical manifestations of functional brain injury, as a result of insult to the head from an external force, e.g., the head being struck by an object, the head striking an object, the head being exposed to forces generated from a blast or explosion, and/or the brain undergoing an acceleration/deceleration movement without direct external trauma to the head with a Glasgow Coma Scale of > 8.

  * The acute, suspected traumatically induced structural brain injury and/or clinical manifestations of functional brain injury will have occurred within the past 24 hours upon admission to the ED.
* The ED normal control group will be males and females ages 18 to 80 (the entire age range), who are admitted to the ED for presenting complaints that do not involve the head or neck (no trauma above the clavicles) and no history of MVA requiring an ED visit or TBI within the past one (1) year, and no primary complaint of syncope

Exclusion Criteria:

* Subjects will be excluded who have forehead, scalp, or skull abnormalities or other conditions that would prevent correct application of the electrode headset on the skin.
* In addition, subjects with dementia, Parkinson's Disease, multiple sclerosis, seizure disorder, brain tumors, history of brain surgery, mentally retarded, psychiatric disorder for which there is a prescribed psychiatric medication taken on a daily basis, substance dependence, history of TIA or stroke within the last year, currently receiving dialysis or in end-stage renal disease, active fever defined as greater than 100oF or 37.7oC, current condition is listed as "critical" in the opinion of the investigator, subject is suffering from an open head injury, subject requires advanced airway management (i.e. mechanical ventilation), currently receiving procedural sedation medications (e.g. benzodiazepine, anesthetic, NMDA receptor antagonist, or opioid agonist), subjects below the age of 18 years, pregnant women, and prisoners will not be eligible for study.
* ED normal control subjects will be excluded if there is a suspected neck injury or trauma above the clavicles, a primary complaint of generalized weakness, or a primary complaint of headache or migraine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who enter the ED at hospitals that are participating as clinical sites for this study
Sampling Method: Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Structural Brain Injury Assessment | within 24 hours of injury
  Using a BrainScope classification algorithm, the Ahead® M-100 will identify subjects showing sensitivities among 3 classes:
  Green - brain electrical activity that is consistent with patients without head injuries (Ahead® M-100 output = 1), Yellow - brain electrical activity that is consistent with head injured subjects who are abnormal, but do not have a structural brain injury (Ahead® M-100 output = 2 or 3), Red - brain electrical activity consistent with a structural brain injury observable on CT (Ahead® M-100 output = 4).

SECONDARY OUTCOMES:
Functional Brain Injury Assessment | within 24 hours of injury
  The sensitivity and specificity to split Yellow from the primary endpoint into two sub groups depending on degree of brain functional impairment observable by an evaluation of the clinical findings on the BrainScope Clinical Charter Patients classified as Yellow (b) will exhibit brain electrical activity consistent with more severe brain functional impairment. Patients classified as Yellow (a) will exhibit brain electrical activity consistent with less severe brain functional impairment observable by an evaluation of the functions on the flow chart.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A De Lorenzo, MD, Principal Investigator — Brooke Army Medical Center; Peter Cuenca, MD, Principal Investigator — Brooke Army Medical Center; Samuel M Galvagno, DO, Principal Investigator — University of Maryland R. Cowley Shock Trauma Center; Stephen J Huff, MD, Principal Investigator — University of Virginia Medical Center; Rosanne Naunheim, MD, Principal Investigator — Washington University - Barnes Jewish Hospital; Brian O'Neil, MD, Principal Investigator — Wayne State University - Detroit Receiving Hospital; Brian J O'Neil, MD, Principal Investigator — Wayne State University - Sinai Grace Hospital; Sandeep Johar, DO, Principal Investigator — Hartford Hospital; Bradley Kolls, MD, Principal Investigator — Duke University Medical Cetner; Jeffrey Bazarian, MD, Principal Investigator — University of Rochester; James Ecklund, MD, Principal Investigator — Inova Fairfax Hospital; Kevin Crutchfield, MD, Principal Investigator — Sinai Hospital
Locations (11):
- United States (11):
  - Hartford Hospital, Hartford, Connecticut
  - University of Maryland R Cowley Shock Trauma Center, Baltimore, Maryland
  - Sinai Hospital, Baltimore, Maryland
  - Wayne State University - Detroit Receiving Hospital, Detroit, Michigan
  - Wayne State University - Sinai Grace Hospital, Detroit, Michigan
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - INOVA Health System, Fairfax, Virginia

REFERENCES:
- [Background] Naunheim RS, Treaster M, English J, Casner T. Automated electroencephalogram identifies abnormalities in the ED. Am J Emerg Med. 2011 Oct;29(8):845-8. doi: 10.1016/j.ajem.2010.03.010. Epub 2010 May 1. PMID 20825903
- [Background] Naunheim RS, Treaster M, English J, Casner T, Chabot R. Use of brain electrical activity to quantify traumatic brain injury in the emergency department. Brain Inj. 2010;24(11):1324-9. doi: 10.3109/02699052.2010.506862. PMID 20722504
- [Background] Naunheim RS, Casner T. Novel method for detecting brain abnormality in a patient with epidural hematoma: a case report. Am J Emerg Med. 2010 Mar;28(3):386.e1-2. doi: 10.1016/j.ajem.2009.05.008. PMID 20223405
- [Background] McCrea M, Prichep L, Powell MR, Chabot R, Barr WB. Acute effects and recovery after sport-related concussion: a neurocognitive and quantitative brain electrical activity study. J Head Trauma Rehabil. 2010 Jul-Aug;25(4):283-92. doi: 10.1097/HTR.0b013e3181e67923. PMID 20611046